CLINICAL TRIAL: NCT02928055
Title: Implanted PNS for Shoulder Pain in Stroke
Brief Title: Peripheral Nerve Stimulation for Shoulder Pain: Dose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Richard Wilson, MD, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB16-00510; R01HD075542 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Shoulder Pain
Keywords: Stroke; Shoulder Pain; Electrical stimulation; Neuromuscular stimulation; Intramuscular stimulation
MeSH Terms: conditions — Stroke; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- PNS (3 hr/day) (Experimental): The PNS (3 hr/day) Group will receive peripheral nerve stimulation treatment for three weeks (3 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period.
  Interventions: Device: Peripheral Nerve Stimulation
- PNS (6 hr/day) (Experimental): The PNS (6 hr/day) Group will receive peripheral nerve stimulation treatment for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period.
  Interventions: Device: Peripheral Nerve Stimulation
- PNS (9 hr/day) (Experimental): The PNS (9 hr/day) Group will receive peripheral nerve stimulation treatment for three weeks (9 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period.
  Interventions: Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad has an embedded power source but also serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for PNS. The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (daily dose is Group-dependent). Stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed. Total time of electrode implantation is no more than 29 days.
  Other Names: Intramuscular Peripheral Nerve Stimulation; Intramuscular Electrical Nerve Stimulation; Smartpatch System

SUMMARY:
The primary objective of this RCT is explore the mechanism for Hemiplegic Shoulder Pain (HSP) reduction due to treatment with peripheral nerve stimulation. We will explore the association of subject-specific clinical and demographic information and pain relief from PNS. We will explore the possible role of central sensitization mechanisms in perpetuating pain via measures of sensory and pain perception. Lastly, we will explore the dose-response association of muscle-contraction from PNS and pain reduction, completion of activities of daily living (ADLs), and improvement in quality of life.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain (HSP) affects up to 60% of moderate to severely impaired stroke survivors. HSP is associated with poor rehabilitation outcomes, including interference with activities of daily living (ADLs) and poor quality of life (QoL). While many treatments for HSP have been proposed, most do not result in long-term relief of pain.

The investigators developed the use of intramuscular peripheral nerve stimulation (PNS) for the treatment of HSP, which involves the temporary placement of a percutaneous intramuscular electrode to stimulate the axillary nerve motor points to the deltoid muscle. The deltoid muscle is stimulated for 6 hours per day for 3 weeks, causing comfortable, non-fatiguing contractions. This treatment, which occurs in the community setting, results in pain relief for up to 12 months when compared to treatment with a hemisling. A systematic review of randomized controlled trials (RCT) with pain as the primary outcome concluded that intramuscular PNS was the only treatment to provide long-term relief of pain for those with HSP. We have completed two RCTs that have demonstrated that a short-term PNS treatment (i.e., 3 or 6 weeks) provides pain relief. The first trial demonstrated efficacy in long-term pain relief in more than 60% of subjects for greater than 12 months. The second trial corroborated the finding that more than 60% of subjects receiving PNS achieved long-term pain reduction, and also showed that PNS reduces pain more than that achieved with physical therapy. The mechanism of action of PNS in reduction of HSP is not yet known. Thus, the primary objective of this RCT is explore the mechanism for HSP reduction.

The mechanisms behind PNS for the treatment of HSP are not known. First, individual variation may contribute to response to PNS, thus we will explore the association of subject-specific clinical and demographic information and pain relief from PNS. Secondly, our team and others have found that in the chronic stage central sensitization mechanisms may also have a role in perpetuating pain, as it does in other forms of chronic shoulder pain. These mechanisms will be explored via measures of sensory and pain perception. Finally, our approach to delivering PNS for HSP is different from other treatments in which PNS is delivered through skin surface electrodes (e.g., transcutaneous electrical nerve stimulation or TENS) in that our treatment produces repeated muscle contraction over the course of weeks. Treatments such as TENS generates tingling sensations (paresthesias) over the painful area, and pain relief following stimulation is short-lived, seldom lasting more than a few hours. We postulate that long-term pain relief for HSP after PNS treatment is due to the repeated muscle contraction that occurs daily over the course of treatment, thus we will explore the dose-response association of muscle-contraction from PNS and pain reduction, completion of activities of daily living (ADLs), and improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain localized to the glenohumeral joint, subacromial area or deltoid insertion associated with: a) rest; b) passive abduction or external rotation range of motion (ROM); c) active abduction ROM; or, d) manual palpation;
* shoulder pain onset or worsening after the most recent stroke;
* weakness of shoulder abductors (≤4/5 on MRC if isolated movement is present);
* ≥ 21-yrs old; < 90-yrs old;
* time of stroke ≥ 3-mo;
* duration of HSP ≥3-mo;
* HSP with moderate to severe pain (BPI SF-3 ≥ 4);
* cognitive and communication ability to fulfill study requirements (cognitive ability based upon a score of ≥24 on the Mini Mental Status Exam (MMSE));
* availability of reliable adult who can assist with study procedures if necessary;
* willing and able to report shoulder pain and other conditions and complete study visits throughout the 4 month study period.

Exclusion Criteria:

* joint or overlying skin infection or history of recurrent skin infections;
* insensate skin;
* need to take > 1 opioid and > 1 nonopioid analgesic medication for HSP;
* regular intake of pain medications for another chronic pain;
* botox injection or subacromial steroid injections to the shoulder within the past 12 wks;
* receiving OT or PT for HSP;
* bleeding disorder or INR > 3.0;
* sensitivity to skin surface electrodes and/or medical-grade adhesives, gels, tapes;
* medical instability;
* pregnancy;
* uncontrolled seizures (>1/mo for 6-mo);
* history of cardiac arrhythmia with hemodynamic instability;
* history of lidocaine allergy;
* history of Parkinson's disease, SCI, TBI, MS, or ipsilateral UE lower motor neuron lesion;
* history of complex regional pain syndrome, myofacial pain syndrome, other pain conditions (investigator discretion);
* cardiac pacemaker or other implanted electronic device;
* history of valvular heart disease (artificial valves, requiring antibiotics for procedures, etc.);
* severely impaired communication.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10; Primary Completion 2019-08 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Wilson, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson RD, Gunzler DD, Bennett ME, Chae J. Peripheral nerve stimulation compared with usual care for pain relief of hemiplegic shoulder pain: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Jan;93(1):17-28. doi: 10.1097/PHM.0000000000000011. PMID 24355994
- [Background] Chae J, Ng A, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Intramuscular electrical stimulation for shoulder pain in hemiplegia: does time from stroke onset predict treatment success? Neurorehabil Neural Repair. 2007 Nov-Dec;21(6):561-7. doi: 10.1177/1545968306298412. Epub 2007 Mar 16. PMID 17369520
- [Background] Chae J, Wilson RD, Bennett ME, Lechman TE, Stager KW. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case series. Pain Pract. 2013 Jan;13(1):59-67. doi: 10.1111/j.1533-2500.2012.00541.x. Epub 2012 Mar 26. PMID 22448759
- [Background] Chae J, Yu D, Walker M. Percutaneous, intramuscular neuromuscular electrical stimulation for the treatment of shoulder subluxation and pain in chronic hemiplegia: a case report. Am J Phys Med Rehabil. 2001 Apr;80(4):296-301. doi: 10.1097/00002060-200104000-00014. PMID 11277137
- [Background] Chae J, Yu DT, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Fang ZP. Intramuscular electrical stimulation for hemiplegic shoulder pain: a 12-month follow-up of a multiple-center, randomized clinical trial. Am J Phys Med Rehabil. 2005 Nov;84(11):832-42. doi: 10.1097/01.phm.0000184154.01880.72. PMID 16244520
- [Background] Wilson RD, Bennett ME, Lechman TE, Stager KW, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case report. Arch Phys Med Rehabil. 2011 May;92(5):837-40. doi: 10.1016/j.apmr.2010.11.003. PMID 21530732
- [Background] Yu DT, Chae J, Walker ME, Fang ZP. Percutaneous intramuscular neuromuscular electric stimulation for the treatment of shoulder subluxation and pain in patients with chronic hemiplegia: a pilot study. Arch Phys Med Rehabil. 2001 Jan;82(1):20-5. doi: 10.1053/apmr.2001.18666. PMID 11239281
- [Background] Yu DT, Chae J, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Feldstein M, Fang ZP. Intramuscular neuromuscular electric stimulation for poststroke shoulder pain: a multicenter randomized clinical trial. Arch Phys Med Rehabil. 2004 May;85(5):695-704. doi: 10.1016/j.apmr.2003.07.015. PMID 15129391
- [Background] Yu DT, Chae J, Walker ME, Hart RL, Petroski GF. Comparing stimulation-induced pain during percutaneous (intramuscular) and transcutaneous neuromuscular electric stimulation for treating shoulder subluxation in hemiplegia. Arch Phys Med Rehabil. 2001 Jun;82(6):756-60. doi: 10.1053/apmr.2001.23310. PMID 11387579
- [Background] Koog YH, Jin SS, Yoon K, Min BI. Interventions for hemiplegic shoulder pain: systematic review of randomised controlled trials. Disabil Rehabil. 2010;32(4):282-91. doi: 10.3109/09638280903127685. PMID 20055567
- [Background] Snels IA, Beckerman H, Lankhorst GJ, Bouter LM. Treatment of hemiplegic shoulder pain in the Netherlands: results of a national survey. Clin Rehabil. 2000 Feb;14(1):20-7. doi: 10.1191/026921500668239146. PMID 10688341
- [Background] Soo Hoo J, Paul T, Chae J, Wilson RD. Central hypersensitivity in chronic hemiplegic shoulder pain. Am J Phys Med Rehabil. 2013 Jan;92(1):1-9; quiz 10-3. doi: 10.1097/PHM.0b013e31827df862. PMID 23255268
- [Background] Wilson RD, Harris MA, Gunzler DD, Bennett ME, Chae J. Percutaneous peripheral nerve stimulation for chronic pain in subacromial impingement syndrome: a case series. Neuromodulation. 2014 Dec;17(8):771-6; discussion 776. doi: 10.1111/ner.12152. Epub 2014 Feb 11. PMID 24512114
- [Background] Wilson RD, Harris MA, Bennett ME, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of shoulder pain from subacromial impingement syndrome. PM R. 2012 Aug;4(8):624-8. doi: 10.1016/j.pmrj.2012.03.002. PMID 22920317
- [Background] Paul TM, Soo Hoo J, Chae J, Wilson RD. Central hypersensitivity in patients with subacromial impingement syndrome. Arch Phys Med Rehabil. 2012 Dec;93(12):2206-9. doi: 10.1016/j.apmr.2012.06.026. Epub 2012 Jul 10. PMID 22789774
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PNS (3 hr/Day) | PNS (6 hr/Day) | PNS (9 hr/Day)
Started | 8 | 8 | 7
End of Treatment | 8 | 8 | 6
1 Month Follow up | 7 | 7 | 6
2 Month Follow up | 6 | 7 | 5
3 Month Follow up | 5 | 6 | 5
Completed (complete study(all milestones)) | 5 | 6 | 5
Not Completed | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PNS (3 hr/Day) | PNS (6 hr/Day) | PNS (9 hr/Day) | Total
Number analyzed (Participants) | 8 | 8 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 4 | 19
  >=65 years | 0 | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.75 (6.25) | 57.5 (8.64) | 62.86 (5.64) | 58.52 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 12
  Male | 3 | 4 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 4 | 2 | 10
  White | 3 | 4 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI)- Short Form (SF) Question 3 (BPI-SF3)
Description: Brief Pain Inventory(BPI) Short Form 3: The BPI has excellent psychometrics and is recommended for the assessment of pain in clinical trials. The developers of the BPI recommend BPI SF-3, the "pain worst" rating, as the primary response metric. The question asks participants to rate their worst pain in the prior 7-d on a 0 to 10 numeric rating scale, where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine." A lower score is better.
Time Frame: End of Treatment (EOT), EOT + 3 mo
Population: numbers analyzed differ at 3 month follow up due to study drop out of some subjects at 3 month follow up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | PNS (3 hr/Day) | PNS (6 hr/Day) | PNS (9 hr/Day)
Number analyzed (Participants) | 8 | 8 | 7
score on a scale
  End of Treatment Score | 5.6 [2 to 9] | 6 [3 to 10] | 5.67 [2 to 9]
  3 month follow up score: number analyzed (Participants) | 5 | 7 | 7
  3 month follow up score | 6.5 [5 to 8] | 5.2 [0 to 10] | 4.4 [3 to 8]

2. Other Pre Specified Outcome: Adverse Events (Related)
Description: Related adverse events are documented as Safety data.
Time Frame: Electrode Implant, Start of Stimulation, 1 week after start of stimulation, 2 weeks after start of stimulation, end of treatment (EOT), EOT + 1mo, EOT + 2 mo, EOT + 3 mo
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: adverse Event were collected for the time frame subject was enrolled in the study. Eligibility through EOT +3 months, an average of 4 months per participant
Arm/Group | PNS (3 hr/Day) | PNS (6 hr/Day) | PNS (9 hr/Day)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNS (3 hr/Day) (N=8) | PNS (6 hr/Day) (N=8) | PNS (9 hr/Day) (N=7)
Fall with injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Fall resulting in avulsion fracture of styloid process
other medical condition: Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) — Reported diagnosis of ca, follow up phase
Orthopedic surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Orthopedic Foot surgery
Anxiety(psychosocial) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Subject hospitalized 2 days for complaints of chest pain after family disagreement. Reported a brief period of suicidal ideation. Discharge diagnosis- chest pain which appeared to be triggered by psychosocial issues
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNS (3 hr/Day) (N=8) | PNS (6 hr/Day) (N=8) | PNS (9 hr/Day) (N=7)
Skin Irritation at Bandage site (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3) | 4 (4) — Itching at bandage site
Skin Irritation under Sprint Pad (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Redness under sprint pad
Retained Lead Fragment (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Lead fragment retained in muscle after explant
Accidental dislodgment of Lead (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 1 (1) — subject accidentally pulled lead out for skin
Fall with injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) — fall with fracture
Skin Irritation at electrode site (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) — redness at electrode site(no infection)
Arm fatigue/weakness/pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) — pain or weakness in shoulder reported after implantation and start of stimulation

LIMITATIONS AND CAVEATS:
The trial did not meet the goal of 10 participants per group. Results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT02928055/Prot_000.pdf